CLINICAL TRIAL: NCT03392454
Title: Measuring the Quality of Life in Patients Receiving a Partial Trapeziectomy (PT) Using a "Minimalist Approach" Versus a Complete Trapeziectomy With Ligament Reconstruction and Tendon Interposition (T+LRTI)
Brief Title: A Case Series Comparing T+LRTI to Partial Trapeziectomy for Thumb Osteoarthritis
Status: Completed | Type: Observational
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Other Study IDs: CMCJ
Record Dates: First submitted 2017-12-06; First posted 2018-01-08 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Arthritis; Health Related Quality of Life; Osteoarthritis
Keywords: Partial Trapeziectomy; Tendon Interposition; Trapeziectomy; Thumb Carpometacarpal Joint
MeSH Terms: conditions — Arthritis; Osteoarthritis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- T+LRTI Patients: Patients who received Trapeziectomy with Ligament Reconstruction and Tendon Interposition.
  Interventions: Procedure: T+LRTI
- PT+TI Patients: Patients who received the Partial Trapeziectomy and Tendon Interposition
  Interventions: Procedure: PT+TI

INTERVENTIONS:
Procedure: T+LRTI — T+LRTI is the most commonly used procedure, it removes the entire trapezium
  Groups: T+LRTI Patients
Procedure: PT+TI — The PT+TI is less invasive than the T+LRTI as only part of the trapezium is removed
  Groups: PT+TI Patients

SUMMARY:
The purpose of this study was to measure the differences in Health Related Quality of Life (HRQOL) and functional measurements between two groups of patients with Carpometacarpal Osteoarthritis of the thumb.

DETAILED DESCRIPTION:
Two patient groups, who have been diagnosed with Carpometacarpal Osteoarthritis of the thumb were compared to measure the Health Related Quality of life (HRQOL) and functional outcomes following two different surgical procedures. The first procedure is currently the most used procedure is North America, Trapeziectomy with Ligament Reconstruction and Tendon Interposition (T+LRTI); this procedure is compared to Partial Trapeziectomy and Tendon Interposition (PT+TI). HRQOL is measured using three questionnaires: one generic, one condition specific and one to measure utility (costs). Patients received their procedures from the respective surgeons and then came in for regular follow up at 1, 3, 6 and 12 months. At these follow up visits the questionnaires and functional measurements (including grip, key pinch and tip pinch strength), were completed

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of advanced stage (Eaton stages II-IV) Carpometacarpal joint (CMCJ) osteoarthritis (OA of the thumb
* Willingness to undergo surgery for CMCJ OA;
* Over the age of 18;
* Able to provide informed consent; and
* Ability to read and comprehend English to complete the HRQOL questionnaires

Exclusion Criteria:

* 1) Diagnosis of Eaton stage I CMCJ OA of the thumb [17]; 2) Under the age of 18; 3) Presence of any concomitant hand pathology (including rheumatoid arthritis, neuropathy and traumatic arthritis); and 4) Previous surgery on the same hand or currently under consideration for other unrelated hand surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (Over the age of 18) who have been diagnosed with CMCJ OA of the thumb, Eaton stages II-IV who are english speaking with no other existing hand pathology.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2012-03-01 (Actual); Primary Completion 2015-11-30 (Actual); Study Completion 2015-11-30 (Actual)

PRIMARY OUTCOMES:
Change in Health Related Quality of Life (HRQOL) as measured by the Short Form 36v2 (SF-36) | 1 week pre-operatively plus 1, 3, 6 and 12 month post-operatively
  The Short-Form 36v2 [SF-36] is a Generic HRQOL questionnaire
Change in Health Related Quality of Life (HRQOL) as measured by the Disabilities of the Arm, Shoulder and Hand (DASH) | 1 week pre-operatively plus 1, 3, 6 and 12 month post-operatively
  The DASH is a condition specific questionnaire
Change in HRQOL as measured by The EuroQol-5D-3L [EQ-5D] | 1 week pre-operatively plus 1, 3, 6 and 12 month post-operatively
  The EQ-5D is a questionnaire that allows utility to be calculated

SECONDARY OUTCOMES:
Change in functional performance as measured by Grip Strength | 1 week pre-operatively and 3, 6 and 12 month post-operatively
  Force applied by the hand, measured by a goniometer in kilograms
Change in functional performance as measured by Two-Point Pinch Strength | 1 week pre-operatively and 1, 3, 6 and 12 month post-operatively
  Force applied by the tip of the thumb and the tip of the index finger, measured by a goniometer in kilograms
Change in functional performance as measured by Key Pinch Strength | 1 week pre-operatively and 3, 6 and 12 month post-operatively
  Force applied by the pad of the thumb and lateral surface of the index finger, measured by a goniometer in kilograms

CONTACTS AND LOCATIONS:
Overall Officials: Achilles Thoma, MD, Principal Investigator — McMaster University

IPD SHARING:
Plan to Share IPD: No
the data will not be made to other researchers, the final results will be anonymized and hopefully published in scientific journals